CLINICAL TRIAL: NCT03498430
Title: An Open Label, Phase I Study of Copanlisib to Evaluate the Pharmacokinetics, Safety and Tolerability in Chinese Patients With Relapsed Indolent Non-Hodgkin's Lymphoma (iNHL)
Brief Title: Copanlisib Chinese PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16866
Record Dates: First submitted 2018-04-08; First posted 2018-04-13 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Indolent Non-Hodgkin's Lymphoma (iNHL) (excluding CLL)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copanlisib (Aliqopa, BAY80-6946) (Experimental): Planned at least 12 patients who meet the entry criteria will receive 60 mg copanlisib as single agent, with dosing on Days 1, 8 and 15 of each 28-day treatment cycle
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (Aliqopa, BAY80-6946) — Copanlisib will be administered intravenously on 60mg once in a 3 weeks-on/1 week-off dose regimen (on Days 1, 8 and 15)

SUMMARY:
This study will be conducted primarily to determine the pharmacokinetics of copanlisib in Chinese patients with relapsed iNHL.

The primary objective of the study is to determine the pharmacokinetics of copanlisib administered on Day1, 8, and 15 of a 28-days cycle (3 weeks-on/1 week off dosing regimen) as a 1 hour intravenous infusion to Chinese patients with relapsed iNHL.

The secondary objectives include the evaluation of safety, tolerability, and tumor response of Chinese patients treated with Copanlisib.

Determine the pharmacokinetics of M-1 metabolite.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and to sign an informed consent form. The informed consent must be signed before any study specific tests or procedures are done
* Chinese, age ≥ 18 years
* Patients with histologically confirmed indolent NHL (excluding chronic lymphocytic leukemia) that have relapsed and who are without past or current central nervous system involvement.
* Patients must have at least 1 measurable lesion according to the Lugano Classification.

  * Patients affected by LPL/WM must have also measurable disease, defined as presence of IgM paraprotein with a minimum IgM level of equal to or greater than 2 times the upper limit of normal (ULN) OR over 10% of lymphoplasmacytic cells in bone marrow.
  * Patients with splenic MZL with splenomegaly but no measurable lesion will be considered eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Prothrombin time (PT) or international normalized ratio (INR) and activated partial thromboplastin time (aPTT) < 1.5 x the upper limit of normal (ULN)
* Adequate bone marrow, liver and renal function
* Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment
* Women of childbearing potential and men must agree to use highly effective contraception from signing of the informed consent form until at least 1 month after the last study drug administration. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control (failure rate of less than 1% per year), e.g. hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence

Exclusion Criteria:

Medical and surgical history:

* Uncontrolled hypertension (Blood pressure ≥ 150/90 mmHg despite optimal medical management)
* Proteinuria of CTCAE grade 3 or higher (> 3.5 g/24 h, measured by urine protein: creatinine ratio on a random urine sample)
* Known bleeding diathesis. Any hemorrhage or bleeding event ≥ Grade 3 within 28 days of start of study medication. (NCI-CTCAE Version 4.03)
* Uncontrolled diabetes with HbA1c ≥ 8.5%
* Ongoing cytomegalovirus (CMV) infection as confirmed by positive polymerase chain reaction (PCR) for CMV

Excluded previous therapies and medications:

* Prior treatment with PI3K inhibitors
* Anticancer chemotherapy or immunotherapy during the study or within 28 days of first study treatment.
* Patients must have recovered from the toxic effects (Grade <2) of the previous anti-cancer chemotherapy or immunotherapy (with the exception of alopecia)
* Biological response modifiers, such as Granulocyte colony stimulating factor (GCSF) within 14 days of first study treatment. G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the principal investigator; however they may not be substituted for a required dose reduction
* Use of strong inhibitors of CYP3A4 is prohibited from Day -14 and for the duration of the study
* Use of St John's Wort or strong inducers of CYP3A4 is prohibited from Day -14 and for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Cmax (Cycle 1 Day 1) of Copanlisib | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start of infusion
  Cmax: maximum observed drug concentration in measured matrix after single dose administration
AUC(0-24) (Cycle 1 Day 1) of Copanlisib | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start of infusion
  AUC: area under the concentration vs. time curve from zero to infinity after single (first) dose
AUC(0-tlast) (Cycle 1 Day 1) of Copanlisib | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start of infusion
Cmax (Cycle 1 Day 15) of Copanlisib | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11 and 24 hours after start of infusion
AUC(0-24) (Cycle 1 Day 15) of Copanlisib | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11 and 24 hours after start of infusion

SECONDARY OUTCOMES:
Overall response rate: proportion of patients with confirmed complete response (CR) and partial response (PR) | Up to about 6 months
Overall disease control rate: proportion of patients who have a best response rating of CR, PR or stable disease (SD) | Up to about 6 months
The number of serious drug-related TEAEs (treatment-emergent adverse events) | Up to about 7 months
The number of non-serious drug-related TEAEs | Up to about 7 months
Cmax (Cycle 1 Day 1) of M-1 metabolite | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start of infusion
AUC(0-24) (Cycle 1 Day 1) of M-1 metabolite | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start of infusion
AUC(0-tlast) (Cycle 1 Day 1) of M-1 metabolite | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start of infusion
Cmax (Cycle 1 Day 15) of M-1 metabolite | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11 and 24 hours after start of infusion
AUC(0-24) (Cycle 1 Day 15) of M-1 metabolite | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11 and 24 hours after start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Beijing Cancer Hospital, Beijing, China

REFERENCES:
- [Derived] Liu W, Ping L, Xie Y, Sun Y, Du T, Niu Y, Cisternas G, Huang F, Garcia-Vargas J, Childs BH, Mehra A, Reschke S, Wang X, Song Y, Zhu J. A phase I pharmacokinetic study of copanlisib in Chinese patients with relapsed indolent non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2022 Jun;89(6):825-831. doi: 10.1007/s00280-022-04417-3. Epub 2022 Mar 23. PMID 35322287
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/